CLINICAL TRIAL: NCT07314684
Title: Impact of GLP1-RAs on Inflammation and Endothelial biomarkerS in Type 2 diABetes meLlitus patiEnts: STABLE-GLP1 Trial
Brief Title: GLP1-RAs Effects on Inflammatory and Endothelial Biomarkers in T2DM
Acronym: STABLE-GLP1
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Pasquale Perrone Filardi, Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2022TF9AH; 2025-520802-37-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-16; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: T2DM (Type 2 Diabetes Mellitus)
Keywords: Type 2 Diabetes Mellitus; Semaglutide; Inflammation; Endothelial function; Biomarkers; Coronary Plaque
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Phase IV low-interventional, Italian, multicenter, randomized, pragmatic clinical trial
Masking Description: Endpoint assessment and statistical analysis will be performed by personnel blinded to treatment assignment to reduce the risk of bias in data interpretation. In addition, the Events Adjudication Committee will be composed of at least three board-certified cardiologists, who are not involved in the conduct of the trial and are blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide in addition to standard therapy (Experimental)
  Interventions: Drug: semaglutide; Drug: Standard Treatment (Guideline-Based)
- Standard therapy alone (Experimental)
  Interventions: Drug: Standard Treatment (Guideline-Based)

INTERVENTIONS:
Drug: semaglutide — The starting dose is 0.25 mg semaglutide once weekly. After 4 weeks the dose should be increased to 0.5 mg once weekly. After at least 4 weeks with a dose of 0.5 mg once weekly, the dose can be increased to 1 mg once weekly to further improve glycaemic control.
  Arms: Semaglutide in addition to standard therapy
Drug: Standard Treatment (Guideline-Based) — Patients will receive standard therapy for T2DM according to standard clinical practice (Guideline-Based). This might include Biguanides, Insulins, Sulfonylureas, SGLT2 inhibitors, Thiazolidinediones, Alpha-glucosidase inhibitors, or DPP-4 inhibitors.

SUMMARY:
Type II diabetes mellitus (T2DM) is a chronic disease associated with a very high risk of developing cardiovascular (CV) events, especially because of its long-term effects. Glucagon-like-peptide-1 receptor agonists (GLP1-RAs) are recommended in subjects suffering from T2DM with a history or at risk for CV disease; however there is a lack of evidence on local actions of GLP1-RAs on inflammation and endothelial function.

The STABLE-GLP1 study aims to evaluate, in patients with T2DM without atherosclerotic cardiovascular disease (ASCVD) or severe target-organ damage (TOD), the possible beneficial effect of semaglutide, a GLP1-AR, on clinical prognosis, inflammatory and endothelial biomarkers.

The STABLE-GLP1 trial is a phase IV interventional, national, multicenter, randomized, pragmatic study, aiming at enrolling 80 patients with T2DM and no ASCVD. Participants will be randomized in 1:1 ratio to receive semaglutide in addition to standard therapy or standard therapy alone, according to body mass index (BMI) category (BMI <30 vs. ≥30 kg/m²). All patients will perform clinical visit, ECG, echocardiography, blood sample collection for endothelial and inflammatory biomarkers dosage at baseline, at 26 weeks, and after 52 weeks of treatment. Data from CTA, performed according to clinical practice before enrollment, will be recorded and retrospectively evaluated to test secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Diagnosis of T2DM in patients without ASCVD or severe TOD but with SCORE2-Diabetes ≥10% with clinical indication in accordance with current guidelines [1] to initiate semaglutide therapy (level of evidence IIa).
* Evaluable, pre-randomization CTA with no evidence of stenosis ≥50% of epicardial coronary vessels, as confirmed by the core laboratory, performed within 2 years prior to inclusion.
* Stable clinical conditions, with controlled blood pressure, lipid profile, and glycemic values, based on assessments performed within 4 weeks prior to inclusion.
* Stable antidiabetic treatment for at least 6 weeks.
* Left ventricular ejection fraction ≥50%.
* For female participants, the participant must not be pregnant or lactating and must be of non-childbearing potential, confirmed at enrollment by one of the following:

  (a) Postmenopausal, defined as amenorrhea for ≥12 months following cessation of fall exogenous hormonal treatments, and with luteinizing hormone and follicle stimulating hormone levels in the postmenopausal range. (b) Documentation of irreversible surgical sterilization by hysterectomy bilateral oophorectomy, or bilateral salpingectomy. Tubal ligation is not considered as irreversible surgical sterilization.
* Ability to understand study procedures and sign informed consent.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Age > 85 years.
* Previous treatment with semaglutide or GLP1-RAs.
* Patients with stenosis of epicardial coronary arteries ≥50%.
* eGFR <45 mL/min/1.73 m2 irrespective of albuminuria or eGFR 45-59 mL/min/1.73 m2 and microalbuminuria (UACR 30-300 mg/g; stage A2) or proteinuria (UACR >300 mg/g; stage A3) or presence of microvascular disease in at least three different sites [e.g. microalbuminuria (stage A2) plus retinopathy plus neuropathy], based on assessments performed within 4 weeks prior to inclusion.
* History of any clinically important disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
* Any history of ASCVD.
* Ongoing New York Heart Association Class IV (heart failure (HF).
* Significant valvulopathy.
* Type 1 diabetes mellitus.
* Hypersensitivity to the active substance or to any of the excipients.
* Known or suspected liver disease, defined by serum transaminase and alkaline phosphatase levels 3 times the normal level.
* Patients with acute inflammatory or infectious diseases during the 3 months prior to inclusion in the study.
* Patients with chronic inflammatory, immune or infectious diseases.
* Patients with a history of cancer within the past 5 years.
* History of alcohol, drug or medication abuse.
* Patients exposed to any other type of radiation, medical or professional.
* Clinically relevant haematological disorders.
* Decompensated metabolic disorders.
* Abuse of alcohol or drugs in the previous 3 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2027-03-08 (Estimated); Study Completion 2027-03-08 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effects of semaglutide in addition to standard therapy on inflammatory biomarkers compared with standard therapy alone in T2DM patients without ASCVD or severe TOD but with SCORE2-Diabetes ≥10%. | From enrollment to the end of treatment at 52 weeks
  Regarding this endpoint, the change in inflammatory biomarkers involved in atherogenesis at follow-up compared to baseline will be evaluated in both treatment arms. Inflammatory biomarkers will be measured in serum using an appropriately validated immunoassay (ELISA - enzyme-linked immunosorbent assay). Inflammatory biomarkers include C-reactive protein (CRP), interleukins (IL-1β, IL-6, IL-10), colony-stimulating factors (M-CSF), tumor necrosis factors (TNF-α), interferons (IFN-γ), transforming growth factors (TGF-β), and adiponectin, all measured in picograms per milliliter (pg/mL).
To evaluate the effects of semaglutide in addition to standard therapy on biomarkers of endothelial dysfunction compared with standard therapy alone in T2DM patients without ASCVD or severe TOD but with SCORE2-Diabetes ≥10%. | From enrollment to the end of treatment at 52 weeks
  Regarding this endpoint, the change in biomarkers involved in endothelial dysfunction at follow-up compared to baseline will be evaluated in both treatment arms. Biomarkers of endothelial dysfunction will be measured in serum using an appropriately validated immunoassay (ELISA - enzyme-linked immunosorbent assay), and include soluble endothelin-1 (ET-1), intercellular adhesion molecule-1 (ICAM-1), vascular cell adhesion molecule-1 (VCAM-1), E-selectin, and P-selectin, all measured in nanograms per milliliter (ng/mL).

SECONDARY OUTCOMES:
To retrospectively evaluate fat attenuation index (FAI) at CTA in T2DM patients without ASCVD or severe TOD but with SCORE2-Diabetes ≥10%. | At baseline retrospectively
  Regarding this endpoint, data from CTA, performed according to clinical practice before enrollment, will be recorded. FAI will be evaluated retrospectively using dedicated software and measured in Hounsfield Units (HU).
To retrospectively evaluate characteristics of subclinical atherosclerotic coronary plaques at CTA in T2DM patients without ASCVD or severe TOD but with SCORE2-Diabetes ≥10%. | At baseline retrospectively
  Regarding this endpoint, data from CTA, performed according to clinical practice before enrollment, will be recorded. Coronary plaque size will be evaluated retrospectively using dedicated software and measured as a percentage (%).
To correlate FAI in T2DM patients without ASCVD or severe TOD but with SCORE2-Diabetes ≥10% to biomarkers evaluated at baseline. | At baseline
  Data from CTA, performed according to clinical practice before enrollment, will be recorded. This outcome measure evaluates the correlation between FAI (measured in Hounsfield Units) at CTA and circulating biomarkers measured at baseline (ng/mL or pg/mL). Correlation will be assessed using Pearson or Spearman correlation coefficients, as appropriate.
To correlate characteristics of subclinical atherosclerotic coronary plaques at CTA in T2DM patients without ASCVD or severe TOD but with SCORE2-Diabetes ≥10% to biomarkers evaluated at baseline. | At baseline
  Data from CTA, performed according to clinical practice before enrollment, will be recorded. This outcome measure evaluates the correlation between coronary plaque size (%) at CTA and circulating biomarkers measured at baseline (ng/mL or pg/mL). Correlation will be assessed using Pearson or Spearman correlation coefficients, as appropriate.
To correlate FAI at CTA to biomarkers evaluated at 52 weeks in T2DM patients without ASCVD or severe TOD but with SCORE2-Diabetes ≥10%. | From enrollment to the end of treatment at 52 weeks
  Data from CTA, performed according to clinical practice before enrollment, will be recorded. This outcome measure evaluates the correlation between FAI (measured in Hounsfield Units) at CTA and circulating biomarkers measured at 52 weeks (ng/mL or pg/mL). Correlation will be assessed using Pearson or Spearman correlation coefficients, as appropriate.
To correlate characteristics of subclinical atherosclerotic coronary plaques at CTA to biomarkers evaluated at 52 weeks in T2DM patients without ASCVD or severe TOD but with SCORE2-Diabetes ≥10%. | From enrollment to the end of treatment at 52 weeks
  Data from CTA, performed according to clinical practice before enrollment, will be recorded. This outcome measure evaluates the correlation between coronary plaque sizes (%) at CTA and circulating biomarkers measured at 52 weeks (ng/mL or pg/mL). Correlation will be assessed using Pearson or Spearman correlation coefficients, as appropriate.
To associate FAI at CTA with the incidence of MACE evaluated at 52 weeks in T2DM patients without ASCVD or severe TOD but with SCORE2-Diabetes ≥10%. | From enrollment to the end of treatment at 52 weeks
  Data from CTA, performed according to clinical practice before enrollment, will be recorded. This outcome measure evaluates the association between FAI (measured in Hounsfield Units) at CTA and the occurrence of major adverse cardiovascular events (MACE) during the follow-up period. MACE will be analyzed as a binary outcome (presence/absence) and reported as incidence (% of patients with at least one event). The association between baseline FAI and MACE will be assessed using logistic regression and/or Cox proportional hazards models (time-to-first event), as appropriate.
To assess the safety of semaglutide in addition to standard therapy compared with standard therapy alone in T2DM patients without ASCVD or severe TOD but with SCORE2-Diabetes ≥10%. | From enrollment to the end of treatment at 52 weeks
  Concerning this endpoint, safety will be measured as the percentage (%) of patients reporting adverse events and/or serious adverse events, and analyzed in both treatment arms.
  An adverse event is any untoward medical occurrence in a patient or clinical study participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse events can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of a medicinal product, whether or not considered drug related.
  A Serious Adverse Event or reaction is any untoward medical occurrence that, at any dose, results in death, is lifethreatening, requires hospitalisation or prolongation of existing hospitalisation, results in persistent or significant disability or incapacity, or is a congenital anomaly or birth defect.
To assess the tolerability of semaglutide in addition to standard therapy compared with standard therapy alone in T2DM patients without ASCVD or severe TOD but with SCORE2-Diabetes ≥10%. | From enrollment to the end of treatment at 52 weeks
  Concerning this endpoint, tolerability will be assessed primarily through treatment discontinuation rates and analyzed in both treatment arms. Discontinuation rates will be measured as the percentage (%) of patients discontinuing treatment.

OTHER OUTCOMES:
To evaluate the effect of semaglutide in addition to standard therapy on time to MACE compared with standard therapy alone in T2DM patients without ASCVD or severe TOD but with SCORE2-Diabetes ≥10%. | From enrollment to the end of treatment at 52 weeks
  Concerning this endpoint, time from randomization to first occurrence of an expanded MACE endpoint consisting of CV death, non-fatal myocardial infarction (MI) (acute MI only), non-fatal stroke (including ischaemic, haemorrhagic and undetermined stroke), unstable angina, or hospitalization for urgent coronary revascularization, will be analyzed in both treatment arms. All events will be determined by an event adjudication committee (EAC).

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Azienda Ospedaliera Sant'Anna e San Sebastiano, Caserta, Caserta
  - Federico II University, Napoli, Napoli

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marx N, Federici M, Schutt K, Muller-Wieland D, Ajjan RA, Antunes MJ, Christodorescu RM, Crawford C, Di Angelantonio E, Eliasson B, Espinola-Klein C, Fauchier L, Halle M, Herrington WG, Kautzky-Willer A, Lambrinou E, Lesiak M, Lettino M, McGuire DK, Mullens W, Rocca B, Sattar N; ESC Scientific Document Group. 2023 ESC Guidelines for the management of cardiovascular disease in patients with diabetes. Eur Heart J. 2023 Oct 14;44(39):4043-4140. doi: 10.1093/eurheartj/ehad192. No abstract available. PMID 37622663